CLINICAL TRIAL: NCT06199245
Title: The Effect of Emotional Freedom Technique on Breastfeeding Success and Self-Efficacy in Primiparous Women in the Early Postpartum Period Who Had a Cesarean Delivery
Brief Title: The Effect of Emotional Freedom Technique on Breastfeeding Success and Self-Efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Eda Yuzuguler, Msc student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IMU-HEM-EY-01
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Breastfeeding; Self Efficacy; Cesarean Delivery Affecting Fetus; First Birth
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: An experimental group in which EFT was applied and a control group in which the routine procedure was applied.
Who Masked: Participant
Masking Description: The researcher knows the distribution of the groups, but the participants do not know whether they are in the experimental or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- emotional freedom technique experimental group (Experimental): Emotional Freedom Technique was applied to the participants in the experimental group, who had a cesarean section on the first postpartum day and agreed to participate in the study, and their breastfeeding self-efficacy and breastfeeding success were evaluated.
  Interventions: Other: emotional freedom technique experimental group
- control group (No Intervention): Participants in the control group were selected from the same sample group, but no intervention was applied. Breastfeeding self-efficacy and breastfeeding success were evaluated after a routine hospital procedure.

INTERVENTIONS:
Other: emotional freedom technique experimental group — Participants in the experimental group, who had a cesarean delivery on the first postpartum day, filled out the sociodemographic and obstetric information form and the Breastfeeding Self-Efficacy Scale, and then were asked to breastfeed their babies and their breastfeeding was evaluated with the Bristol Breastfeeding Evaluation Scale. The participant was then asked to score her breastfeeding between 0 and 10 to evaluate her Subjective Units of Disturbance Scala (SUD) score. The next evaluation was made 2 hours after the participant received breastfeeding training, the Bristol Breastfeeding Rating Scale score was obtained, and the SUD was scored again after 2 rounds of Emotional Freedom Techniques (EFT) application. Finally, at the end of the day, 2 rounds of EFT application were performed by taking the SUD score before the EFT session, and after the application, the participant's Breastfeeding Self-Efficacy Scale, Bristol Breastfeeding Evaluation Scale and SUD scores were recorded.
  Arms: emotional freedom technique experimental group

SUMMARY:
This study was planned to determine the effect of emotional freedom technique (EFT) on breastfeeding success and self-efficacy in primiparous women in the early postpartum period who had a cesarean delivery.

DETAILED DESCRIPTION:
Breast milk is an easily digestible, natural food that reduces the morbidity and mortality of the newborn and contains the fluid, energy and nutrients necessary for its physical, spiritual and mental development. Breastfeeding not only has a biological effect on the mother and baby, but also has an emotional effect and has many immunological, psychological, social and economic benefits for both mother and baby. Therefore, it is of great importance that the baby be fed exclusively with breast milk for the first 6 months and that breastfeeding continues until the age of 2.

EFT, a needle-free and emotional form of acupuncture, is an energy technique that emerged from the idea that "The cause of all negative emotions is the disruption in the body's energy system." EFT; It can be safely applied to individuals of all ages, including the elderly, pregnant women and children. When looking at the literature, no studies were found regarding breastfeeding and EFT. It has been observed that primiparous women, especially those who have had a cesarean section, have difficulty breastfeeding. It is thought that breastfeeding will be reinforced and improved with EFT, which helps to eliminate negative emotions in the subconscious and create a positive mood.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35,
* Primiparous and giving birth by cesarean section,
* Having a spontaneous pregnancy,
* Wound, scar, infection etc. in the tapping area. without conditions,
* Women who do not have verbal communication problems

Exclusion Criteria:

* Being outside the age range of 18-35
* Has any problem that prevents communication,
* Those who gave birth normally
* Having had a high-risk pregnancy,
* Women who want to leave the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study is conducted with women who have given birth by cesarean section.
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Bristol Breastfeeding Rating Scale | one day
  This scale measures breastfeeding success. The scale is a Likert-type scale consisting of 4 items: "positioning", "holding", "sucking" and "swallowing". Each item is scored between 0-2 points. The lowest score from the scale is 0, the highest score is 8. Low scores indicate that breastfeeding is not effective, while high scores indicate that breastfeeding is effective.

SECONDARY OUTCOMES:
breastfeeding self-efficacy scale | one day
  This scale measures breastfeeding self-efficacy. The scale is a 5-point Likert type scale. The minimum score that can be obtained from the scale is 14, the maximum score is 70, and the scale has no cut-off point.
Subjective Units of Disturbance Scala | one day
  This scale is used in energy therapies and evaluates the individual's discomfort. The scale is scored between 0 and 10, where "0" means no discomfort and "10" means unbearable discomfort and is scored between 0 and 10. As the number value increases, the discomfort experienced by the person becomes more severe.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar IRMAK VURAL, Asst. Prof., Study Director — thesis advisor
Locations (1):
- Medipol Mega University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No